CLINICAL TRIAL: NCT00803660
Title: In Practice Survey on the Treatment of Hypertension in Patients With Type 2 Diabetes.
Brief Title: Survey on the Treatment of Hypertension in Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Vo Viet Tuan, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CVN-DUM-2008/1
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-07

CONDITIONS: Hypertension; Type 2 Diabetes
Keywords: hypertension; BP; diabetes; anti-hypertensive treatment; ACE-I; ARB
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Multi-centre survey of type 2 diabetic patients who are currently on anti-hypertensive treatment. Data collection for each patient will take place at one visit. To observe the proportion of diabetic patients on antihypertensive treatment reaching the BP<130/80 mmHg. To observe the proportion of diabetic patients on antihypertensive treatment reaching the BP<130/80 mmHg by treatment groups. To observe the proportion of patients achieving a therapeutic glycemic response defined as HbA1c=<7%. To observe the proportion of patients achieving fasting plasma glucose<110 mg%. To identify factors for not achieving BP<130/80 mmHg. To describe percentage of patients with positive proteinuria (including microalbuminuria) by treatment groups .

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Patient was diagnosed with type 2 diabetes
* Patient is on antihypertensive treatments for at least 3 months, with the same regimen for a minimum of 4 weeks prior to survey

Exclusion Criteria:

* Patients are critically ill, had mental health problems or difficulty in communication
* Patients who are unwilling or unable to provide informed consent
* Involvement in the planning and conduct of the study (applies to both AstraZeneca staff or staff at the study site).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 diabetic patients who are currently using antihypertensive treatment for at least 3 months, with same regimen for a minimum of 4 weeks prior to the survey
Sampling Method: Probability Sample
Enrollment: 1060 (Estimated)
Dates: Start 2008-11; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The number of patients achieving the BP<130/80 mmHg
The percentage of patients achieving the BP<130/80 mmHg

SECONDARY OUTCOMES:
The number and percentage of patients achieving the BP<130/80 mmHg by treatment groups
The number and percentage of patients achieving HbA1c=<7%
The number and percentage of patients achieving the FPG<110 mg%
The association between unachievement of BP<130/80 mmHg and other factors (age, gender, CV risk factors, CV and diabetes history, duration of type of treatment...)
The number and percentage of patients with positive proteinuria by treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Dang Van Phuoc, PhD., Principal Investigator — University of Medicine and Pharmacy of HCMC; Pham Nguyen Vinh, PhD., Principal Investigator — Tam Duc Heart Hospital; Pham Gia Khai, PhD., Principal Investigator — Vietnam Heart Association; Nguyen Thy Khue, PhD, Principal Investigator — Endocrinology and Diabetes Association of HCMC
Locations (19):
- Vietnam (19):
  - Research Site, Châu Đốc, An Giang
  - Research Site, Bạc Liêu, Bac Lieu
  - Research Site, Qui Nhon, Binh Dinh
  - Research Site, Cà Mau, Ca Mau
  - Research Site, Can Tho, Can Tho City
  - Research Site, Da Nang, Da Nang
  - Research Site, Buon Me Thuoc, Dak Lak
  - Research Site, Biên Hòa, Dong Nai
  - Research Site, Thống Nhất, Dong Nai
  - Research Site, Dong Thap, Dong Thap
  - Research Site, Hanoi, Hanoi
  - Research Site, Nha Trang, Khanh Hoa
  - Research Site, Kiến Giang, Kien Giang
  - Research Site, Nam Định, Nam Dinh
  - Research Site, Thái Bình, Thai Binh
  - Research Site, Huế, Thua Thien
  - Research Site, Tiền Giang, Tien Giang
  - Research Site, Haiphong
  - Research Site, Ho Chi Minh City